CLINICAL TRIAL: NCT07097337
Title: Point of Care Fibrinogen Measurement in Trauma Patients in the Emergency Department
Acronym: POCFIB
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Diagnostica Stago R&D (Industry)
Responsible Party: Principal Investigator, Niki Ottenhof, Dr., Erasmus Medical Center
Other Study IDs: POCFIB
Record Dates: First submitted 2025-06-12; First posted 2025-07-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Trauma Induced Coagulopathy; Trauma Coagulopathy; Fibrinogen Deficiency; Fibrinogen; Deficiency, Acquired; Massive Transfusion Protocol; Massive Hemorrhage
Keywords: point of care fibrinogen; trauma induced coagulopathy; fibrinogen suppletion; fibrinogen
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients for which the massive transfusion protocol is activated and transfusion is initiated

SUMMARY:
Background: Why This Study Matters When someone suffers a severe injury (like from a car crash), they can bleed heavily. One complication doctors often face is something called Trauma-Induced Coagulopathy (TIC). This is a condition where the blood doesn't clot properly, making bleeding worse. The reasons behind TIC are complicated and not fully understood.

One important substance involved is fibrinogen, a protein that helps blood clot. Low levels of fibrinogen are often the first sign of TIC and tend to be linked with how bad the injury is. Because of this, doctors have been giving trauma patients extra fibrinogen early on, hoping it will help them survive.

However, a recent large study (called CRYOSTAT-2) showed that giving high doses of fibrinogen to all trauma patients didn't actually help reduce deaths. This suggests that not everyone needs it-only patients with very low fibrinogen levels (below 1.5 grams per liter) should get it.

The problem is: it currently takes 30 to 45 minutes to get fibrinogen test results. In emergency situations, that's too slow. So doctors have been guessing who needs it, which might not always be the best approach.

What This Study Aims to Do This new study wants to see if a faster, bedside test-called a point-of-care (POC) fibrinogen test-can be used in the Emergency Department (ED) during trauma resuscitations.

Main Goals:

Feasibility: Can the test be done quickly and easily during emergency care?

Usefulness: If the fast test had been available, would doctors have made different decisions-like giving or not giving fibrinogen? And would that have changed outcomes for the patients?

Study Details Feasibility Study: To see if the test is practical during trauma care.

Retrospective Cohort Study: To look back at patients and see if early test results could have changed decisions or outcomes.

Who's In the Study? Adults over 16 who arrive at the ED with serious trauma and for whom the hospital's Massive Transfusion Protocol was activated (meaning they had major bleeding).

They must have received at least one unit of blood.

How the Study Will Work The Test: A small amount of blood (0.15 ml) will be taken from blood that's already being drawn for routine care-so no extra blood draws are needed.

The POC test (called qLabs Fib) will be done at the same time as standard lab tests.

Important Note: Doctors won't make decisions based on this fast test for now. It's just being tested for feasibility.

Nurses will note how long the test takes and if they had any trouble using it.

Later, researchers will look back at the data to see:

* What the fibrinogen levels were.
* Whether the fast results could have helped guide better treatment.
* If outcomes like how much blood was given or survival were affected.

Why It Matters If the fast test works well, it could lead to

* Faster, more accurate treatment in trauma cases.
* Less unnecessary use of fibrinogen, saving resources and avoiding possible side effects.
* Better outcomes for patients by tailoring treatment to their actual needs.

DETAILED DESCRIPTION:
Rationale:

Worldwide, trauma accounts for 5.8 million deaths every year and trauma is the leading cause of death under the age of 44. Up to 25% of trauma victims have clotting abnormalities known as trauma induced coagulopathy (TIC). TIC is a complex, multifactorial coagulation disorder of which the exact pathophysiology is not completely understood. Patients with TIC have a three- to four-fold increased risk of death. While many factors have been identified to influence TIC, fibrinogen is thought to be one of the central players. A low level of fibrinogen is one of the first signs of TIC and there is a strong relation between fibrinogen levels and injury severity.

Measuring fibrinogen levels in the clinical laboratory takes a long time (30-45min), therefore fibrinogen suppletion in acute massive hemorrhage is usually empirical. Several observational studies showed clinical benefit from fibrinogen suppletion in trauma. However, the CRYOSTAT-2 trial, a multi-center randomized controlled trial, did not find a mortality benefit for empirical treatment with high dose fibrinogen.

Trauma patients presented at the emergency department (ED) are currently treated using an integrated approach commonly known as damage control resuscitation. The focus of treatment is 1. Identify and stop ongoing bleeding, and 2. Hemostatic resuscitation consisting of supplementing the blood loss by red blood cell, plasma, and platelet transfusion in prespecified ratios. Coagulation correction by administration of tranexamic acid, calcium and fibrinogen is often included in massive transfusion protocols. As soon as laboratory results become available, the empirical treatment transfers into goal directed treatment based on the lab results. Until now it has been impossible to use a goal directed approach for coagulation correcting in the first hour after arrival in the ED because results from coagulation tests take 30-45min to become available.

In summary, fibrinogen plays an important role in TIC and a low fibrinogen is related to worse outcomes, however, empirical treatment with fibrinogen in the trauma patient suspected of massive hemorrhage does not lead to improved outcomes. A goal directed approach based on real time fibrinogen measurements would therefore be preferred.

This study was initiated because recently a point of care (POC) fibrinogen test was introduced, making a fast determination of fibrinogen values possible. Stago BNL introduced the qLabs FIB Monitoring system. This POC analyzer can measure fibrinogen levels within 1-10 minutes. The lower the fibrinogen level, the quicker the result. Clinically relevant levels of fibrinogen (<2g/l) are available within 2-3 minutes. The use of this POC fibrinogen measurement could result in a goal directed suppletion of fibrinogen and could potentially improve coagulation and outcomes. Because the use of a POC fibrinogen test is new, the current study is initiated to determine if using a POC fibrinogen test is feasible in the ED. Moreover, the study will determine if POC fibrinogen testing could potentially alter the current practice of fibrinogen suppletion by retrospective analysis of the fibrinogen values, fibrinogen suppletion, transfusion strategy and clinical outcomes.

Objective(s) For this study, point of care (POC) fibrinogen measurements will be introduced in the emergency department (ED). The main objective will be to determine feasibility of POC fibrinogen measurements in the ED during trauma resuscitation. Moreover, the study will retrospectively evaluate if the fibrinogen values would have resulted in different clinical decisions on fibrinogen suppletion if they were available to the treating team and if this could have influenced clinical outcomes.

Study type Feasibility study and retrospective cohort study

Study population Adult trauma patients will be identified as follows: (1) by the trauma team leader on admission to the ED or (2) by the research team personnel following a massive transfusion protocol activation. Patients will be assessed for eligibility to enter the trial according to the criteria set out below. If patients are eligible for entry into the study following initial screening, they will be enrolled automatically under deferred consent. Patients will be considered eligible for enrolment in this trial if they fulfil all the inclusion criteria and none of the exclusion criteria detailed below.

Inclusion criteria

To be eligible to participate in this study, a subject must meet the following criteria:

* The participant is judged to be an adult (according to the attending clinician, e.g. 16 years or older) and has sustained traumatic injury
* The participant is deemed by the attending clinician to have on-going active hemorrhage
* The major hemorrhage protocol (MTP) is activated or this patient and transfusion is initiated

Exclusion criteria

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* The participant has been transferred from another hospital
* The trauma team leader deems the injuries incompatible with life

Methods When a patient is presented at the emergency department who meets the inclusion criteria and none of the exclusion criteria, the patient is included in the study.

Because the MTP has been activated and transfusion has been initiated, standard clinical care dictates that blood is drawn, including a 2.7ml citrate tube (BD vacutainer citrate tube) which is used for conventional coagulation testing. An ER nurse takes the citrate tube to the room where blood gas analysis is performed. Once the blood gas sample is loaded into the machine, the ER nurse will perform the POC fibrinogen testing as described in the user manual8.

To perform the POC fibrinogen test, 0,15ml is removed from the citrate tube (BD vacutainer citrate tube). Removing 0.15ml does not influence the integrity of the sample or the ability to perform the usual analysis on the sample. No additional blood will be drawn for this testing. The 0,15ml citrated blood is then loaded into the cartridge of the qLabs FIB monitoring system. The sample is tested. The ER nurse is instructed not to wait for the test results to become available. He/she will confirm that the test has started and then resume the normal clinical tasks. The results from the measurement will be saved on the qLabs FIB monitoring meter and collected at a later stage by a member of the research team for analysis. The result will not be made available for the treating team and will not be recorded in the electronic patient file. No clinical decisions will be made based on this measurement.

For each POC fibrinogen measurement the nurse will be asked to report the time it took to perform the test, whether the measurement was eventful and whether difficulties arose. This will be documented in the log provided in the ER. The nurse will be asked to complete this information after the patient has left the ER or the nurse is no longer needed for patient care.

Burden and risks The burden and the risks are very low in this study. Standard of care will not be influenced by this study. No additional blood sampling or any other additional procedures will be performed. Patients will not be asked to fill in questionnaires or participate actively in the research. The clinical outcome data will be anonymized and stored on a data platform with the highest level of security, keeping the risks as low as possible.

To perform the POC fibrinogen test a nurse will be occupied for a few minutes. During these minutes the nurse would otherwise be available for clinical tasks. To limit this amount of time, the nurses will be trained to efficiently perform the measurement. Moreover, the POC fibrinogen measurement will be performed alongside the blood gas analysis, which normally takes the nurse of the floor for a few minutes. Therefore, the burden and risks of this study will remain minimal.

Recruitment and consent All participants will be enrolled in the study without informed participant consent due to the emergency nature of the trial (i.e. a "deferred consent" will be applied). The research team will monitor the ongoing status of the participants and their ability to provide informed consent. If the participant does not regain capacity, a personal and/or professional consultee's advice is sufficient for the participant to remain in the study for the ongoing collection of follow-up data. When a participant regains capacity to give consent, full information will be provided to them, and they will be asked to sign a consent form agreeing to their continuation in the study.

Analysis Data will be analyzed with the Statistical Package for the Social Sciences (SPSS) version 29 or higher (SPSS, Chicago, II., USA). Normality of continuous variables will be tested with Shapiro-Wilk test, homogeneity in variance with the Levene's test.

Descriptive analysis will be performed to rapport the data. For continuous data the mean with SD (parametric data) or the median with percentiles (non-parametric data) will be calculated. For categorical data percentages will be calculated.

Privacy protection The pseudonymized database will be stored on a workspace of the DRE, for the duration of the study. Only researchers involved in the study will be granted access to the DRE through their personal log in. Data security will be guaranteed by using the DRE, which has the highest level of security in data handling. After completion of the study, the data will be permanently stored on the Research Storage. All servers provided by the Erasmus MC IT department.

The handling of personal data will comply with the EU General Data Protection Regulation and the Dutch Act on Implementation of the General Data Protection Regulation (in Dutch: Algemene Verordening Gegevensbescherming en Uitvoeringswet Algemene Verordening Gegevensbescherming).

ELIGIBILITY:
Population (base) Adult trauma patients will be identified as follows: (1) by the trauma team leader on admission to the ED or (2) by the research team personnel following a massive transfusion protocol activation. Patients will be assessed for eligibility to enter the trial according to the criteria set out below. If patients are eligible for entry into the study following initial screening, they will be enrolled automatically under deferred consent. Patients will be considered eligible for enrolment in this trial if they fulfil all the inclusion criteria and none of the exclusion criteria detailed below.

Inclusion criteria

To be eligible to participate in this study, a subject must meet the following criteria:

* The participant is judged to be an adult (according to the attending clinician, e.g. 16 years or older) and has sustained traumatic injury
* The participant is deemed by the attending clinician to have on-going active hemorrhage
* The major hemorrhage protocol (MTP) is activated or this patient and transfusion is initiated

Exclusion criteria

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* The participant has been transferred from another hospital
* The trauma team leader deems the injuries incompatible with life

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients for which the massive transfusion protocol has been activated and transfusion has been initiated.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of qLabs Fib testing in the emergency department | 2 hours after inclusion
  Feasibility of qLabs Fib testing in the ED, where feasibility will be determined by percentage of qLabs Fib results available within 30min after patient arrival in the ED.

SECONDARY OUTCOMES:
Incidents during testing | 2 hours after inclusion
  For all POC fibrinogen measurements it will be recorded if there were problems with the test (percentage of test without problems) and if so what problems occurred.
Total number of transfusion products uses | 24 hours
  Units of erythrocytes, plasma and thrombocytes will be recorded for the first 24hours after trauma
6hr, 24hr and 30d mortality | 30 days
  Percentage of mortality will be recorded at 3 different time points
Coagulation measurements in the first 24hrs | 24 hours
  Prothrombin Time (PT) (seconds, normal range 10-13), Activated Partial Thromboplastin Time (APTT) (seconds, normal range 25-40), International Normalized Ratio (INR) (, and Fibrinogen levels between 1.5-4.5 g/L. will be measured directly after arrival at the ED and when indicated during the first 24h after trauma
Trauma mechanism | 2 hours after inclusion
  Trauma mechanism will be recorded. This includes blunt trauma (e.g., falls, vehicle collisions), penetrating trauma (e.g., gunshot or stab wounds), and thermal or chemical injuries.
Injury severity score | 2 hours after inclusion
  Injury severity score will be calculated and recorded as descibed below:
  Each injury is categorized using the AIS, a scale from 1 (minor) to 6 (unsurvivable).
  Body Regions:
  Injuries are categorized into six body regions: Head and Neck, Face, Chest, Abdomen, Extremities (including pelvis), and External.
  ISS Calculation:
  Identify the highest AIS score for each of the six body regions. Select the three highest AIS scores from different body regions. Square each of these three scores. Sum the squared values to get the ISS.
  Interpretation:
  The ISS correlates with mortality, morbidity, and hospital stay. An ISS > 15 is commonly used as a threshold for defining major trauma.
  Major Trauma:
  Defined by an ISS greater than 15.
  Unsurvivable Injury:
  If any injury is assigned an AIS of 6, the ISS is automatically assigned a value of 75,
Blood pressure on ED presentation | 2 hours after inclusion
  Blood pressure will be recorded on ED presentation (mmHg)
Pulse on ED presentation | 2 hours after inclusion
  Pulse will be recorded on ED presentation (beats/minute)
Respiratory rate on ED presentation | 2 hours after inclusion
  Respiratory rate will be recorded on ED presentation (breaths/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline van der Marel, MD, PhD, Study Director — Erasmus Medical Center; Niki A. Ottenhof, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White NJ. Mechanisms of trauma-induced coagulopathy. Hematology Am Soc Hematol Educ Program. 2013;2013:660-3. doi: 10.1182/asheducation-2013.1.660. PMID 24319248